CLINICAL TRIAL: NCT00290186
Title: An Evaluation of the Therapeutic Effectiveness of Hyperbaric Oxygen Treatments and Hyperbaric Air Treatments for Children With Cerebral Palsy
Brief Title: An Evaluation of Hyperbaric Treatments for Children With Cerebral Palsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated for futility.
Sponsor: Dayton Children's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03038007; FWP20020014H; DAMD17-03-2-0060; HSRRB-12213; CMC 04-024; KMCN 03-021
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spastic Cerebral Palsy; CP; Hyperbaric; HBOT
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric Oxygen Treatment (HBO) (Experimental): 100% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  Interventions: Device: Hyperbaric Oxygen Treatment
- Hyperbaric Air Treatment (HBA) (Active Comparator): 14% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  Interventions: Device: Hyperbaric Air Treatment

INTERVENTIONS:
Device: Hyperbaric Oxygen Treatment — 100% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  Other Names: HBOT; HBO
  Arms: Hyperbaric Oxygen Treatment (HBO)
Device: Hyperbaric Air Treatment — 14% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  Other Names: HBAT; HBA
  Arms: Hyperbaric Air Treatment (HBA)

SUMMARY:
The study is to evaluate the effectiveness of hyperbaric treatments and the potential longer-term effects in children between the ages of 3 and 8 years with spastic cerebral palsy (CP). One group will receive 100% oxygen and the other group will receive the equivalent of 21% oxygen (room air). The children will receive pre-treatment testing (baseline). After 40 experimental treatments are completed, the children will be retested at 0, 3, and 6 months to evaluate any changes.

DETAILED DESCRIPTION:
The study proposed herein is a randomized, double blind study to evaluate the therapeutic effectiveness of HBO in children (ages 3-8 years) with a diagnosis of spastic CP. Ninety-four children will be randomly assigned to either a hyperbaric oxygen treatment group or hyperbaric air treatment (HBA) group. Each group will receive 40 dives of 60 minutes duration each at 1.5 atmospheres of pressure (ATA) (the HBO group receiving 100% oxygen, and the HBA group receiving an air mixture containing 14% oxygen, which simulates 21% oxygen at 1.5 ATA).

Neurological testing (Gross Motor Function Measure, Pediatric Evaluation of Disability Inventory, and the Test of Variables of Attention) will be performed at baseline, immediately after experimental treatment #40, and at 3 and 6 months after experimental treatment #40. Statistical analysis will be performed on these test data to determine any changes from baseline, or between group differences, in the functional capabilities of the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children, ages 3 to 8 years with a diagnosis of spastic cerebral palsy.
* No documented evidence of hypoxic-ischemic encephalopathy (HIE). Hypoxic-ischemic encephalopathy (HIE) is not one of the major causes of CP.
* Medically cleared to participate. Your child's primary care physician will be asked to medically clear your child before entering the study.
* Able to pass pretest screening exercise. Each child will undergo the following screening exercise to determine the likelihood of being able to participate in the study: In order to assess ability to tolerate the placement of the oxygen hood in the hyperbaric setting, a hyperbaric oxygen hood will be placed upon the shoulders, or body of your child (depending upon size of your child) and with encouragement and comforting by you and study nurse, the child will be asked to maintain the placement of the hood for 15 minutes. Each child will be asked to blow through a straw, blow the nose, drink through a straw, or to swallow on command.

Exclusion Criteria:

* Any previous HBO treatments.
* Thoracic surgery within 6 months of beginning the study.
* Unstable epilepsy as determined by a history of having had more than one major motor (generalized or partial tonic/clonic) seizure within the past six months. Having multiple motor seizures, requiring more than three anticonvulsant drugs for seizure control; or requiring changes in seizure medications more than once per month.
* Significant pulmonary dysfunction as determined by a history of chronic pulmonary disease, cystic fibrosis, interstitial lung disease, or chronic shortness of breath or cough. Uncontrolled asthma/reactive airway disease.
* Significant behavioral problems requiring medication.
* Any major congenital deformities of the brain or spinal cord.
* Active pneumothorax (collapsed lung).
* Recent cancer treatment with cisplatinum, bleomycin, or doxorubicin.
* Certain heart problems that cause the heart to pump poorly as determined by a history of congenital heart disease, cardiomyopathy, or symptoms of chest pain, dizziness, and shortness of breath.
* Optic neuritis.
* Diabetics requiring insulin therapy.
* Spherocytosis.
* Major GI reflux with frequent emesis.
* Botulinum toxin A (Botox) treatments within 6 months of entering study.
* Before entering the study, we will require that chronic medications be unchanged for the prior three months except for minor dosage adjustments.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2005-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lacey, MD, PhD, Principal Investigator — Children's Medical Center of Dayton, Neurologist
Locations (2):
- United States (2):
  - Dayton Children's Hospital, Dayton, Ohio
  - Wound Healing and Hyperbaric Medicine Center, Wpafb, Ohio

REFERENCES:
- [Result] Lacey DJ, Stolfi A, Pilati LE. Effects of hyperbaric oxygen on motor function in children with cerebral palsy. Ann Neurol. 2012 Nov;72(5):695-703. doi: 10.1002/ana.23681. Epub 2012 Oct 15. PMID 23071074

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyperbaric Oxygen Treatment (HBO): Hyperbaric Oxygen Treatment: 100% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  25 Were allocated to HBO 24 Completed all 40 treatments
  1 Withdrawn during treatments due to right ear problems and rectal bleeding 24 Completed post treatment testing
  1. Study terminated prior to 3-month followup testing
  2. Did not return for 3- or 6-month followup testing
  1 Missed 3-month followup due to illness not related to study but returned for 6-month followup testing 20 Completed 3-month followup testing 20 Completed 6-month testing 24 Included in pre and post treatment analyses 20 Included in pre, post, and 3-month analyses 20 Included in pre, post, 3-month and 6-month analyses
- Hyperbaric Air Treatment (HBA): Hyperbaric Air Treatment: 14% oxygen at 1.5 ATA for 60 mins, Mon-Fri, 40 treatments total
  24 Were allocated to HBA 22 Completed all 40 treatments
  1 Withdrew prior to treatments
  1 Withdrawn during treatments for seizures due to shunt malfunction 22 Completed post treatment testing
  1 Study terminated prior to 3-month followup testing 21 Completed 3-month followup testing
  1 Did not return for 6-month followup testing
  1 Missed 6-month followup testing due to illness not related to study 19 Completed 6-month followup testing 22 Included in pre and post treatment analyses 21 Included in pre, post, and 3-month analyses 19 Included in pre, post, 3-month and 6-month analyses
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Started | 25 | 24
Completed Baseline Assessments | 25 | 24
Completed 8 Weeks of Treatment | 24 | 22
Completed Post-treatment Assessments | 24 | 22
Completed 3-month Followup Assessments | 20 | 21
Completed 6-month Followup Assessments | 20 | 19
Completed | 20 | 19
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Study was terminated prior to 3-month te | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA) | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 24 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (1.3) | 5.2 (2.0) | 5.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Gross Motor Function Classification System (GMFCS) level [Number; unit: participants] — GMFCS© Robert Palisano, Peter Rosenbaum, Stephen Walter, Dianne Russell, Ellen Wood, Barbara Galuppi, 1997. CanChild Centre for Childhood Disability Research, McMaster University. (Reference: Dev Med Child Neurol 1997;39:214-223).
  Levels I-V based on self-initiated movement, with emphasis on sitting, transfers, and mobility. Level I is highest functioning, level V is lowest
  General:
  I: walks without limitations II: walks with limitations III: walks using hand-held mobility device IV: self-mobility with limitations; may use powered mobility V: transported in manual wheelchair
  participants
    I | 6 | 4 | 10
    II | 1 | 1 | 2
    III | 2 | 4 | 6
    IV | 3 | 6 | 9
    V | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Total Score (GMFM-88).
Description: GMFM-88: total percent score on 88 items (I) of motor function grouped into 5 dimensions: A) lying and rolling (17 I), B) sitting (20 I), C) crawling and kneeling (14 I), D) standing (13 I), E) walking, running, jumping (24 I). Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Scores in each dimension determined by dividing score obtained by maximum possible score for that dimension, and multiplying by 100. Range is 0-100% for each: the higher the percent score, the greater the functional ability.
  Dimension scores and total GMFM-88 score calculated as:
  A) lying and rolling: (score achieved/51)x100 B) sitting: (score achieved/60)x100 C) crawling and kneeling: (score achieved/42)x100 D) standing: (score achieved/39)x100 E) walking, running, and jumping: (score achieved/72)x 100 GMFM-88 = (%A+%B+%C+%D+%E)/number of dimensions GMFM-66: [(total score on subset of 66 items/198)x100]
Time Frame: Baseline (within 1 week of starting 8-week treatment period) and post-treatment (within 1 week of ending 8-week treatment period)
Population: Analysis included all participants who completed baseline assessments (within 1-week of start of treatment), 40 hyperbaric treatments, and post-treatment assessments (within 1 week of ending treatment).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 1.5 [-0.3 to 3.3] | 0.6 [-1.0 to 2.2]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.539, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI [-1.5 to 3.3]

2. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure 66-Item Subscale Score (GMFM-66).
Description: GMFM-66: total percent score on 66-item subscale of GMFM-88: Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score determined by dividing score obtained by maximum possible score for the 66 items, and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. GMFM-66: [(total score on subset of 66 items/198)x100].
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 1.2 [-0.1 to 2.2] | 1.1 [-0.1 to 2.4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.921, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.6 to 1.8]

3. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Dimension A
Description: Total percent score on 17 items of GMFM grouped into Dimension A) lying and rolling. Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score in Dimension A determined by dividing score obtained by maximum possible score for that dimension (51), and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. A) lying and rolling: (score achieved/51)x100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 1.1 [-1.3 to 3.6] | 0.1 [-3.3 to 3.5]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.945, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-3.0 to 5.1]

4. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Dimension B
Description: Total percent score on 20 items of GMFM grouped into Dimension B) sitting. Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score in Dimension B determined by dividing score obtained by maximum possible score for that dimension (60), and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. B) sitting: (score achieved/60)x100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | -0.1 [-2.3 to 2.1] | 1.4 [-1.7 to 4.4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.342, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.1 to 2.2]

5. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Dimension C
Description: Total percent score on 14 items of GMFM grouped into Dimension C) crawling and kneeling. Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score in Dimension C determined by dividing score obtained by maximum possible score for that dimension (42), and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. C) crawling and kneeling: (score achieved/42)x100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 3.0 [-1.0 to 6.9] | -0.5 [-4.0 to 2.9]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.149, ANCOVA; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-1.6 to 8.6]

6. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Dimension D
Description: Total percent score on 13 items of GMFM grouped into Dimension D) standing. Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score in Dimension D determined by dividing score obtained by maximum possible score for that dimension (39), and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. D) standing: (score achieved/51)x100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 1.7 [-1.7 to 5.1] | 0.7 [-1.5 to 2.9]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.685, ANCOVA; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-3.0 to 5.1]

7. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Score (Post-treatment Minus Pre-treatment) on Gross Motor Function Measure Dimension E
Description: Total percent score on 24 items of GMFM grouped into Dimension E) walking, running, and jumping. Each item scored on 0-3 scale: 0 = does not initiate, 1 = initiates, 2 = partially completes, 3 = completes. Score in Dimension E determined by dividing score obtained by maximum possible score for that dimension (72), and multiplying by 100. Range is 0-100%: the higher the percent score, the greater the functional ability. E) walking, running, and jumping: (score achieved/72)x 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 1.6 [-0.6 to 3.8] | 1.3 [-0.3 to 2.8]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.584, ANCOVA; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.4 to 3.0]

8. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Functional Skills: Self-care
Description: Primary caregiver-reported (through structured interview) child capabilities for 73 items of functional skills grouped under self-care. Scores are 0 = unable to perform; 1 = capable of performing. Scores range from 0-73 and are rescaled to a 0-100% scale. Higher scores indicate greater abilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 4.4 [2.3 to 6.5] | 3.3 [1.6 to 5.0]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.498, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-1.5 to 3.7]

9. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Functional Skills: Mobility
Description: Primary caregiver-reported (through structured interview) child capabilities for 59 items of functional skills grouped under mobility. Scores are 0 = unable to perform; 1 = capable of performing. Scores range from 0-59 and are rescaled to a 0-100% scale. Higher scores indicate greater abilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 2.8 [1.2 to 4.4] | 2.7 [0.7 to 4.6]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.945, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.3 to 2.2]

10. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Functional Skills: Social Function
Description: Primary caregiver-reported (through structured interview) child capabilities for 65 items of functional skills grouped under social function. Scores are 0 = unable to perform; 1 = capable of performing. Scores range from 0-65 and are rescaled to a 0-100% scale. Higher scores indicate greater abilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 2.1 [0.4 to 3.8] | 1.9 [0.4 to 3.4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.932, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.1 to 2.4]

11. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Caregiver Assistance: Self-care
Description: Primary caregiver-reported (through structured interview) amount of caregiver assistance required by child to complete 8 items of daily activity grouped under self-care. Scores are 0 = total assistance, 1 = maximal assistance, 3 = minimal assistance, 4 = supervise/prompt/monitor, 5 = independent. Total scores range from 0-40 and are rescaled to 0-100%. Higher scores indicate greater ability to perform independently.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 4.9 [2.8 to 6.9] | 2.6 [1.3 to 3.9]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.051, ANCOVA; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-0.2 to 4.7]

12. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Caregiver Assistance: Mobility
Description: Primary caregiver-reported (through structured interview) amount of caregiver assistance required by child to complete 7 items of daily activity grouped under mobilityare. Scores are 0 = total assistance, 1 = maximal assistance, 3 = minimal assistance, 4 = supervise/prompt/monitor, 5 = independent. Total scores range from 0-35 and are rescaled to 0-100%. Higher scores indicate greater ability to perform independently.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 2.7 [-0.1 to 5.6] | 3.4 [1.5 to 5.2]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.648, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.0 to 2.8]

13. Secondary Outcome: The Difference Between Groups (HBO Minus HBA) in Change in Scores (Post-treatment Minus Pre-treatment) on Pediatric Evaluation of Disability Inventory (PEDI) Caregiver Assistance: Social Function
Description: Primary caregiver-reported (through structured interview) amount of caregiver assistance required by child to complete 5 items of daily activity grouped under social function. Scores are 0 = total assistance, 1 = maximal assistance, 3 = minimal assistance, 4 = supervise/prompt/monitor, 5 = independent. Total scores range from 0-25 and are rescaled to 0-100%. Higher scores indicate greater ability to perform independently.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 24 | 22
units on a scale | 0.7 [-1.7 to 3.1] | 2.4 [0.4 to 4.4]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.473, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.7 to 1.4]

14. Secondary Outcome: The Difference Between Groups in Change in Scores (Post-treatment Minus Pre-treatment) on the Test of Variables of Attention (TOVA): Number of Correct Responses.
Description: One of 4 parts of the TOVA, a computerized continuous performance test that measures attention and impulsivity in visual mode. Measures the number of times a target is correctly selected when it appears on a screen. Score ranges from 0-160; higher scores represent greater number of correct responses.
Time Frame: as for outcome 1
Population: The TOVA was only administered to patients who were 4-8 years old, not visually impaired, and able to complete a practice test. Analysis included all eligible participants who completed baseline assessments (within 1-week of start of treatment), 40 hyperbaric treatments, and post-treatment assessments (within 1 week of ending treatment).
Measure: Mean (95% Confidence Interval); unit: number of correct responses
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 7 | 3
number of correct responses | 12 [-22 to 46] | -34 [-175 to 108]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.157, t-test, 2 sided; Mean Difference (Final Values) = 46, 95% CI 2-sided [-22 to 114]

15. Secondary Outcome: The Difference Between Groups in Change in Scores (Post-treatment Minus Pre-treatment) on the Test of Variables of Attention (TOVA): Number of Correct Nonresponses.
Description: One of 4 parts of the TOVA, a computerized continuous performance test that measures attention and impulsivity in visual mode. Measures the number of times a target is correctly not selected (number of times a child correctly refrains from hitting a buzzer) when it appears on a screen. Score ranges from 0-160; higher scores represent greater number of correct nonresponses.
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: Number of correct nonresponses
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 7 | 3
Number of correct nonresponses | 3 [-6 to 12] | 4 [-6 to 14]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: positive values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.876, t-test, 2 sided; Mean Difference (Final Values) = -1, 95% CI 2-sided [-15 to 13]

16. Secondary Outcome: The Difference Between Groups in Change in Scores (Post-treatment Minus Pre-treatment) on the Test of Variables of Attention (TOVA): Response Time in Milliseconds
Description: One of 4 parts of the TOVA, a computerized continuous performance test that measures attention and impulsivity in visual mode. Measures the processing time in milliseconds that it takes to correctly respond to a target. Lower times represent better response times. Range = 0 - 2000 milliseconds
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: time in milliseconds
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 7 | 3
time in milliseconds | -45 [-113 to 23] | 33 [-164 to 231]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: negative values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.167, t-test, 2 sided; Mean Difference (Final Values) = -79, 95% CI 2-sided [-198 to 41]

17. Secondary Outcome: The Difference Between Groups in Change in Scores (Post-treatment Minus Pre-treatment) on the Test of Variables of Attention (TOVA): Response Time Variability in Milliseconds
Description: One of 4 parts of the TOVA, a computerized continuous performance test that measures attention and impulsivity in visual mode. Measures the variability in processing time in milliseconds that it takes to correctly respond to a target. Response time variability = the standard deviation of response times for correct responses. Lower values represent less variability and better responses. Range of response times = 0-2000 milliseconds.
Time Frame: as for outcome 1
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: time in milliseconds
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Number analyzed (Participants) | 7 | 3
time in milliseconds | -47 [-110 to 15] | -9 [-220 to 201]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Treatment (HBO) vs Hyperbaric Air Treatment (HBA); Between-group difference: negative values represent greater improvement in HBO group; Test type: Superiority or Other; p = 0.468, t-test, 2 sided; Mean Difference (Final Values) = -38, 95% CI 2-sided [-153 to 77]

ADVERSE EVENTS:
Arm/Group | Hyperbaric Oxygen Treatment (HBO) | Hyperbaric Air Treatment (HBA)
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/24
Other Adverse Events (participants affected / at risk) | 7/25 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (HBO) (N=25) | Hyperbaric Air Treatment (HBA) (N=24)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
fluid in ear and nose (Ear and labyrinth disorders) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (HBO) (N=25) | Hyperbaric Air Treatment (HBA) (N=24)
ear pain (Ear and labyrinth disorders) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes